CLINICAL TRIAL: NCT07085156
Title: The Efficacy and Safety of Reduced-Intensity Conditioning With Fludarabine- Melphalan-Busulfan for Allogeneic Hematopoietic Stem Cell Transplantation in the Treatment of Myelodysplastic Syndromes
Brief Title: Reduced Intensity Conditioning for MDS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Wuhan TongJi Hospital (Other); Wuhan Children's Hospital (Wuhan Maternal and Child Healthcare Hospital), Tongji Medical College, Huazhong University of Science and Technology (Unknown); Zhejiang University (Other)
Responsible Party: Principal Investigator, Hu Xiaoxia, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-BMT-012
Record Dates: First submitted 2025-07-06; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: MDS
Keywords: MDS; Reduced intensity conditioning
MeSH Terms: interventions — fludarabine; Melphalan; Busulfan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FBM arm (Experimental): Adult MDS patients eligible for allo-HCT will receive Fludarabine 30mg/m^2 d-6 to -2; melphalan 70mg/m^2 d-6; busulfan 3.2mg/kg d-4 to -3 as conditioning regimen.
  Interventions: Drug: Fludarabine; melphalan; busulfan

INTERVENTIONS:
Drug: Fludarabine; melphalan; busulfan — The conditioning regimen includes fludarabine, busulfan, and melphalan, with a transplant conditioning intensity of 3.0. The RIC is used in the allo-HCT in the MDS patients.

SUMMARY:
Allogeneic hematopoietic cell transplantation (allo-HCT) is the only potential cure for Myelodysplastic syndrome (MDS). Currently, the conditioning regimen for MDS allogeneic transplantation still follows AML, and there are fewer explorations in this field. In a large-scale retrospective analysis with 532 MDS undergoing allo-HCT, reduced intensity conditioning is resulted in improved overall survival (OS), reduced non-relapse mortality (NRM) , while sparing relapse.

Therefore, the investigators conduct a prospective, single-arm, multicentre study to evaluate the efficacy and safety of Fludarabine-Melphalan-Busulfan reduced-intensity conditioning in MDS patients.

DETAILED DESCRIPTION:
This study is a prospective, multicenterstudy designed to evaluate the efficacy and safety of evaluate the efficacy and safety of Fludarabine-Melphalan-Busulfan intermediate-intensity transplantation conditioning regimen for the treatment of MDS. . Patients with MDS who are eligible for enrolment were pretreated with a Fludarabine-Melphalan-Busulfan regimen (Fludarabine 30mg/m2d-6 to -2; melphalan 70mg/m2d-6; busulfan 3.2mg/kg d-4 to -3). The primary endpoint is 2-year relapse-free survival (RFS) after transplantation. Secondary endpoints includes 2-year post-transplant survival (OS) and cumulative recurrence rate at 2 years post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-70 (including boundaries) and gender;
* Diagnosis of MDS is confirmed on the basis of bone marrow cytomorphology, immunophenotyping and chromosomal and molecular biology tests;
* IPSS-R intermediate-risk or higher-risk or IPSS-M intermediate-risk or higher-risk MDS; transfusion-dependent MDS;
* ECOG score≤ 3 points;
* Have appropriate organ function, and laboratory results within 7 days prior to the start of trial treatment need to meet the following criteria:
* Aspartate aminotransferase (AST) ≤ 3 times ULN (upper limit of normal, ULN);
* Alanine aminotransferase (ALT) ≤ 3x ULN;
* Total serum bilirubin ≤ 1.5 times the upper limit of normal ULN unless the patient has documented Gilbert syndrome; patients with Gilbert-Meulengracht syndrome with bilirubin ≤ 3.0 times the upper limit of normal and direct bilirubin ≤ 1.5 times the upper limit of normal may be included;
* Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60 mL/min;
* Coagulation function: International Normalised Ratio (INR) ≤ 1.5 x ULN, Activated Partial Thromboplastin Time (APTT) ≤ 1.5 x ULN;
* Left ventricular ejection fraction (LVEF) ≥50%;
* Voluntarily signing the informed consent, understanding and complying with the requirements of the study, good compliance, and cooperating with the follow-up visits.

Exclusion Criteria:

* Allergies or contraindications to any of the drugs in the protocol;
* Currently have clinically significant active cardiovascular disease such as uncontrolled arrhythmias, uncontrolled hypertension, congestive heart failure, any grade 3 or 4 heart disease as determined by the New York Heart Association (NYHA) functional class, or a history of myocardial infarction within the 6 months prior to screening;
* Serious medical conditions that may limit the patient's participation in this trial (e.g., progressive infection, uncontrolled diabetes);
* Active autoimmune diseases such as SLE, rheumatoid arthritis, etc;
* Patients with neurological or psychiatric disorders;
* The patient is pregnant or breastfeeding;
* Those who are unable to understand or comply with the study protocol or are unable to sign the informed consent form.
* Other conditions that, in the opinion of the investigator, make the patient otherwise unsuitable for participation in this study;

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
2-year relapse-free survival after transplantation | through study completion, an average of 2 year
  relapse

SECONDARY OUTCOMES:
2-year post-transplant survival | through study completion, an average of 2 year
  survival
Cumulative recurrence rate at 2 years post-transplant | through study completion, an average of 2 year
  relapse

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China